CLINICAL TRIAL: NCT05849220
Title: Dapagliflozin in Non Alcoholic Fatty Liver Disease Associated Cirrhosis and Its Role in Preventing Development of Chronic Kidney Disease. A Randomized Controlled Trial.
Brief Title: Dapagliflozin in Non Alcoholic Fatty Liver Disease Associated Cirrhosis and Its Role in Preventing Development of Chronic Kidney Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-57
Record Dates: First submitted 2023-03-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-03

CONDITIONS: NAFLD Cirrhosis
MeSH Terms: interventions — dapagliflozin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin+Standard of Care (Experimental): Dapagliflozin
  Interventions: Drug: Dapagliflozin; Other: Standard of Care
- Standard of Care (Active Comparator): Standard of Care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin
  Arms: Dapagliflozin+Standard of Care
Other: Standard of Care — Standard of Care

SUMMARY:
The role of Dapagliflozin in the improvement in CKD in both diabetic and non-diabetic patients has been evaluated in the past. SGLT2i have also been found to be beneficial in NAFLD patients in improving the liver function parameters. It is also known that cirrhotic patients are at a higher risk of developing CKD at 1 year when compared to non cirrhotics. With this study we aim to study the role Dapagliflozin in cirrhotic patients in reducing the development of CKD, its impact on cirrhotic cardiomyopathy and its role in improvement of metabolic profile and liver related outcomes.

DETAILED DESCRIPTION:
Hypothesis: Investigator hypothesise that Use of Dapagliflozin in NAFLD-Cirrhotic patients with moderate ascites will prevent progression and development of chronic kidney disease, ameliorate metabolic dysfunction and facilitate resolution of ascites by its renoprotective, cardioprotective and metabolic effects

Aim: To evaluate the efficacy of Dapagliflozin in NAFLD-cirrhotic patients with moderate ascites in preventing progression and development of CKD

Methodology:

Study population:

* Age > 18 years <70 years
* Patient with NAFLD associated cirrhosis and moderate ascites
* Stable eGFR-(>60 ml/min/1.73m2) calculated using MDRD-6 equation: eGFR (ml/min/1.73 m2) = 198 × [serum creatinine (mg/dL)]-0. 858 × [age]-0. 167 × [0.822 if patient is female] × [serum urea nitrogen concentration (mg/dL)]-0.

Study design: Monocentric open label randomised controlled study. The study will be conducted in Department of Hepatology, ILBS.

Study period: 1 year

Sample size: Based on the previous study, assuming that progression rate in standard arm for chronic kidney disease is 30% and with addition of Dapagliflozin Investigator expect that there will be an absolute reduction of 20% in progression, i.e. 10 % progression rate

* Alpha - 5%
* Power - 80
* 10 % dropout rate
* Investigator need to enrol approximately 144 patients with 72 patients in each arm allocated into two groups by block randomization method taking block size of 10.

Patients will be evaluated in OPD for stable eGFR (based on the creatinine value in the last 3 months)

Intervention Patients after screening for all exclusion criteria will be randomised into 2 arms (group-1, receiving Dapagliflozin) and (group-2, standard of care) in a ratio 1:1

Monitoring and assessment Both the groups will undergo baseline investigations including KFT, Urine routine and microscopy, LFT, Fibroscan liver and spleen, baseline 2decho, ECG, NTproBNP, biomarkers of inflammation, renal reserve and metabolic profile incuding Hba1c, FBS, S.lipid profile, waist circumference, HOMA-IR, BMI, Bone mineral density(DEXA), liver frailty index, 6 min walk test and hand grip analysis.

All the patients will be followed in OPD at 3 monthly intervals and biomarkers of renal reserve and inflammation will be repeated at 6 monthly interval.

STATISTICAL ANALYSIS: Continuous data- Student's t test

* Nonparametric analysis- Mann Whitney test
* Survival outcome By Kaplan-Meier method curve.
* For all tests, p≤ 0.05 will be considered statistically significant.
* Analysis will be performed using SPSS.
* The analysis will be done with intention to treat and per protocol analysis if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years <70years
* Patient with NAFLD associated cirrhosis and moderate ascites
* Stable eGFR-(>60 ml/min/1.73m2) calculated using MDRD-6 equation: eGFR (ml/min/1.73 m2) = 198 × [serum creatinine (mg/dL)]-0. 858 × [age]-0. 167 × [0.822 if patient is female] × [serum urea nitrogen concentration (mg/dL)]-0.
* Valid Informed written consent

Exclusion Criteria:

* Hospitalized patients
* CTP-C patients
* Intrinsic/structural kidney disease, obstructive uropathy, ADPKD, Anatomic urologic defects that predispose to urinary tract infection
* History of organ transplantation
* Refractory Ascites
* Type 1 DM
* History of hypoglycemic symptoms in the last 2 months
* Recurrent UTI
* Patient with HCC or portal vein thrombosis
* Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor
* History of fracture in the preceding year
* Severe Hyponatremia (Na <125 MEq/L)
* Pregnancy or Lactating mother
* Receiving cytotoxic therapy, immunosuppressive therapy or other immunotherapy for primary or secondary renal disease within 6 months prior to enrolment
* MI, unstable angina, stroke or transient ischemic attack (TIA) within 12 weeks prior to enrolment
* Coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG]) or valvular repair/replacement within 12 weeks prior to enrolment or is planned to undergo any of these procedures after randomization
* Mixed ascites (additional etiology of ascites apart from portal hypertension)
* Any severe extra hepatic condition including respiratory and cardiac failure
* Acute-on-chronic liver failure as per the APASL criteria
* Refusal to give consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants developing Chronic Kidney Disease at 1 yr defined as per KDIGO guidelines. | 1 year

SECONDARY OUTCOMES:
Number of participants developing Chronic Kidney Disease. | 3 months
Number of participants developing Chronic Kidney Disease. | 6 months
Improvement in eGlomerular filtration rate (eGFR) at 3 months. | 3 months
Change in eGlomerular filtration rate (eGFR) at 6 months. | 6 months
Change in eGlomerular filtration rate (eGFR) at 12 months. | 12 months
Number of participants developing acute kidney disease at 3 months. | 3 months
Number of participants developing acute kidney disease at 6 months. | 6 months
Number of participants developing acute kidney disease at 12 months. | 12 months
Number of participants Discontinuing drug due to adverse effects. | 1 year
Number of participants with resolution of ascites - partial or complete at 3 months. | 3 months
Number of participants with resolution of ascites - partial or complete at 6 months. | 6 months
Number of participants with resolution of ascites - partial or complete at 12 months. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided